CLINICAL TRIAL: NCT04059692
Title: Immediate Effect of a Single Cervical Spinal Manipulation on Cervical Movement Pattern
Brief Title: Immediate Effect of a Single Cervical Spinal Manipulation
Acronym: SMCervical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID0025
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Neck Pain
Keywords: neck pain; manual therapy; movement
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: The study design is experimental
Who Masked: Participant, Outcomes Assessor
Masking Description: The subjects do not know the group to which they belong. The evaluator does not know the treatment applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical manipulation intervention (Experimental): To perform the evaluation and detect the cervical vertebral level with mobility restriction, with the patient in supine position, a cervical examination is carried out to determine the mobility restriction, both in flexo-extension, as in inclination and rotation. To check the level of restriction, the post-anterior sliding test is performed.
  The manipulation is performed following the criteria of thrust manipulations. A maximum of 3 manipulations are applied in total per subject, one for each level (high level C1-C2, medium level C3-C6, and low level C7), if necessary.
  Interventions: Other: Placebo intervention
- Placebo intervention (Placebo Comparator): This group will receive 15 minutes of sham techniques in a supine position over the stretcher. First, a series of short-time and no pressure contact with physiotherapist´s hands is performed in several points of head and shoulders for 10 minutes. Subsequently, light touch is applied on standardized anatomic areas, for 2 minutes each time.
  Interventions: Other: Cervical manipulation intervention

INTERVENTIONS:
Other: Cervical manipulation intervention — Cervical manipulative technique
  Arms: Placebo intervention
Other: Placebo intervention — Sham intervention
  Arms: Cervical manipulation intervention

SUMMARY:
Objective: The aim of the present study is to analyze the immediate effect of a single cervical spinal manipulation on cervical movement pattern. Further, To perform the sample size calculation, the investigators took into consideration that the investigators pretend to achieve a medium effect size (d=0.5) of the differences with two groups (EG and CG) and two aimed to explore the impact on pain, disability and patient's improvement-perceived sensation, comparing with a placebo.

Methods: The study design is experimental and purposive sampling was used to select the study participants. The grouping allocation was randomized. The people volunteer to participate in the study, are assigned to the experimental group (EG) that will receive a single manipulation, to the control group (CG) that will receive a single placebo treatment.

The participants will be assessed twice, one before the treatment and the other, after the end. Head movement is recorded by means of a video-photogrammetry system from the coordinates of a set of eight reflective markers located on a helmet. The movements will be record at 200 fps.

In each evaluation, the perceived pain and the neck disability index are also recorded. And the impression of change is evaluated only in the second evaluation.

Outcomes. Pain, Disability of the neck, Impression of Change, Range of motion (RoM), Maximum angular velocity (MAV), Maximum angular acceleration (MAA) and Harmonicity (HARM).

Intervention: The intervention, in both groups, it includes only one session that lasted 15 minutes approximately: a) Cervical manipulation intervention and b)Placebo intervention.

DETAILED DESCRIPTION:
INTRODUCTION Non-specific neck pain is defined as pain in the posterior and lateral aspect of the neck between the superior nuchal line and the spinous process of the first thoracic vertebra with no signs or symptoms of major structural pathology. It is a common musculoskeletal disorder that leads to substantial disability, discomfort, and reduced cervical mobility, resulting in enormous health costs in terms of treatment and work absenteeism. The American Physical Therapy Association's guidelines on neck pain recommends utilizing cervical manipulation (CM) and mobilization procedures to reduce neck pain based on strong evidence. Spinal manipulation is defined as "a passive, high velocity, low amplitude thrust applied to a joint complex within its anatomical limit with the intent to restore optimal motion, function, and/or to reduce pain" and its effectiveness, concretely of a continuous program of cervical manipulations (CM), on neck pain has been largely studied. A previous systematic review concluded that treatments based on CM are effective both alone and in combination with exercises whilst other systematic reviews and an evidence-based guideline showed that CM, combined with exercises, resulted to be more effective for neck pain, function, and global perceived effect, than a therapeutic program based, exclusively, on CM.

Nevertheless, the underlying mechanisms of the pain decrease with this therapeutic approach are not completely understood. A recent study aimed at analyzing the biomechanics of a single CM, used a complex system of synchronized biplane radiographs to measure the facet gapping during a single manipulation. Authors demonstrated that target and adjacent motion segments undergo facet joint gapping during a manipulation and that segmental and global range of motion (ROM) increases in all three planes of motion immediately after one manipulation.

In the clinical setting, the best of our knowledge, only one previous clinical trial have analyzed the effectiveness of a single cervical manipulation on cervical range of motion, comparing with placebo, demonstrating an improvement in all the global maximum cervical movements, measured with the goniometer. However, pain may affect other movement' characteristics beside the maximum range of motion (ROM), as velocity, variability or movement harmony.

Nevertheless, no previous study has analyzed the characteristics of the patients' cervical motion pattern after a single manipulation which could provide information about functional changes in cervical movements. People with neck pain, has shown more slow movements, less harmonic movements in the points close to pain and exponential trend at the ends of the range, even when cervical spine motion ranges remain within normal limits.

The investigators hypothesized that functional assessment of the cervical spine based on the analysis of the motion pattern, will let us know if a single manipulation is effective in the improvement of those variables.

The aim of the present study is to analyze the immediate effect of a single cervical spinal manipulation on cervical movement pattern. Further, the investigators aimed to explore the impact on pain, disability and patient's improvement-perceived sensation, comparing with a placebo.

METHODS Participants The study design is experimental and purposive sampling was used to select the study participants. The grouping allocation was randomized. The people volunteer to participate in the study, are assigned to the experimental group (EG) that will receive a single CM, to the control group (CG) that will receive a single placebo treatment.

All the participants should meet the following inclusion criteria: perceived pain scored 3 or above, in a visual analogue scale, and neck functional status revealing a mild disability. Additionally, patients had symptoms duration less than 30 days.

For both groups, the exclusion criteria include an inflammatory rheumatic disease or an inner ear disorder, the use of antidepressant opioid or sedative drugs, current vertigo or dizziness, visual loss, neurological disorder, and trunk or shoulder surgery within the past year.

Sample size To perform the sample size calculation, the investigators took into consideration to achieve a medium effect size (d=0.5) of the differences with two groups (EG and CG) and two assessments (pre and post-treatment). Further, the investigators set a type I error of 5%, and a type II error of 20%. This power calculation resulted in 17 patients on each group.

Assessment procedures The participants will be assessed twice, one before the treatment and the other, after the end. Head movement is recorded by means of a video-photogrammetry system from the coordinates of a set of eight reflective markers located on a helmet. The movements will be record at 200 fps.

Participants sit in a chair with the trunk fixed at the back by means of belts. In each session, they perform three movements: flexion-extension (FE), lateral flexion (LB) and axial rotation (AR) whose order was randomized. Each movement will be perform seven consecutive times without stopping and achieving a continuous and smooth cyclic movement with the maximum achievable range at their preferred speed. The participants are encouraged to practice the three movements before the test begins, to avoid the learning effect.

In each evaluation, the perceived pain and the neck disability index are also recorded. And the impression of change is evaluated only in the second evaluation.

Outcomes Pain, with the Visual Analogue Scale (VAS), in which the patients marked their level of pain intensity on a 10-cm horizontal line (0= no pain to 10= maximum pain) at the time the assessment was carried out.

Disability of the neck, with the 'Neck Disability Index', a self-report questionnaire used to determine how neck pain affects a patient's daily life. Scoring is reported on a 0-50 scale, 0 being the best possible score.

Impression of Change, with the self-reported measure 'Patient Global Impression of Change' that reflects a patient's belief about the efficacy of treatment.

Range of motion (RoM): angular excursion of the cervical motion. Maximum angular velocity(MAV), it is measured as percentile 95 of angular velocity during the test.

Maximum angular acceleration(MAA), it is measas percentile 95 of angular acceleration during the test.

Harmonicity (HARM): is the absolute value of the correlation coefficient between two motion. Thus HARM quantifies the fit between the actual movement and the simple harmonic motion.

Intervention The intervention, in both groups, it includes only one session that lasted 15 minutes approximately. Participants should wear a sleeveless shirt that allows the physiotherapist to treat the neck region. Evaluations and manipulations are performed by the same experienced physiotherapist.

Cervical manipulation intervention Prior to intervention, a screened for any signs of vertebrobasilar insufficiency is performed by means of the vertebral artery compromise test, as well as the root compression test using the Jackson test, and the screening for upper cervical spine ligamentous instability through Sharp-Purser test, alar ligament stress test and transverse ligament test.

To perform the evaluation and detect the cervical vertebral level with mobility restriction, with the patient in supine position, a cervical examination is carried out to determine the mobility restriction, both in flexo-extension, as in inclination and rotation. To check the level of restriction, the post-anterior sliding test is performed.

Once the vertebral levels with restriction have been detected, high speed and low amplitude manipulation is carried out based on the location of the pain and the detection of the perceived joint hypomobility, using the clinical criterion for this, with a maximum of 2 manipulative attempts by vertebral level, regardless of having achieved joint cavitation. The manipulation is performed following the criteria of thrust manipulations. A maximum of 3 manipulations are applied in total per subject, one for each level (high level C1-C2, medium level C3-C6, and low level C7), if necessary.

Placebo intervention This group will receive 15 minutes of sham techniques in a supine position over the stretcher. First, a series of short-time and no pressure contact with physiotherapist´s hands is performed in several points of head and shoulders for 10 minutes. Subsequently, light touch is applied on standardized anatomic areas, equal to those treated with manipulative intervention, for 2 minutes each time, adding a total duration of approximately 15 minutes, similar to the intervention group.

Statistics Standard statistical methods will be use to obtain the mean and standard deviation of the mean (SD). For the inferential analysis of the data, a mixed two-factor multivariate analysis of variance (MANOVA) with a between-subject factor 'group' (i.e. CG and EG) ant a within-subject factor 'time' with two groups (pre and post-intervention). Multiple comparison techniques are performed using Bonferroni correction. The investigators will evaluate the assumption of homoscedasticity and it will be assumed in each variable. In addition, the investigators will compare the perceived changes after treatment between the two groups with an independent Student T test. Type I error will be set as <5% (p <.05).

ELIGIBILITY:
Inclusion Criteria:

* Perceived pain scored 3 or above, in a visual analogue scale
* Neck functional status revealing a mild disability
* Minimun duration of the symptoms being one month.

Exclusion Criteria:

* inflammatory rheumatic disease or an inner ear disorder.
* the use of antidepressant opioid or sedative drugs.
* current vertigo or dizziness.
* visual loss.
* neurological disorder,
* trunk or shoulder surgery within the past year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Range of motion | 1 day
  Angular excursion of the cervical motion.
Harmonicity | 1 day
  Is the absolute value of the correlation coefficient between: Ӫ and Ө. Thus Harmonicity quantifies the fit between the actual movement and the simple harmonic motion.

SECONDARY OUTCOMES:
Disability of the neck | 1 day
  To determine how neck pain affects a patient's daily life. Scoring is reported on a 0-50 scale, 0 being the best possible score.
Impression of Change | 1 day
  The self-reported measure 'Patient Global Impression of Change' that reflects a patient's belief about the efficacy of treatment. This is a one-item questionnaire in which patients rank their change following an intervention on a scale from 1 to 7 (1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; 7, very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí-López, Principal Investigator — Faculty of Physiotherapy. University of Valencia
Locations (1):
- Gemma Victoria Espí-López, Valencia, Spain

REFERENCES:
- [Result] Rey-Eiriz G, Alburquerque-Sendin F, Barrera-Mellado I, Martin-Vallejo FJ, Fernandez-de-las-Penas C. Validity of the posterior-anterior middle cervical spine gliding test for the examination of intervertebral joint hypomobility in mechanical neck pain. J Manipulative Physiol Ther. 2010 May;33(4):279-85. doi: 10.1016/j.jmpt.2010.03.005. PMID 20534314
- [Result] Puentedura EJ, Landers MR, Cleland JA, Mintken PE, Huijbregts P, Fernandez-de-Las-Penas C. Thoracic spine thrust manipulation versus cervical spine thrust manipulation in patients with acute neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2011 Apr;41(4):208-20. doi: 10.2519/jospt.2011.3640. Epub 2011 Feb 18. PMID 21335931
- [Derived] Serra-Ano P, Venegas W, Page A, Ingles de la Torre M, Aguilar-Rodriguez M, Espi-Lopez G. Immediate Effects of a Single Session of Cervical Spine Manipulation on Cervical Movement Patterns in People With Nonspecific Neck Pain: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2023 Jan;46(1):17-26. doi: 10.1016/j.jmpt.2023.05.006. Epub 2023 Jul 7. PMID 37422751